CLINICAL TRIAL: NCT05917665
Title: Early Digital, Analyte and Neurologic Biomarkers of Acute and Chronic Brain Injury and Recovery in CQT Instructors
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Leslie Saxon, MD, Professor of Medicine, Executive Director, USC Center for Body Computing,, University of Southern California
Other Study IDs: Brain Health CQT
Record Dates: First submitted 2023-05-10; First posted 2023-06-26 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; mTBI; concussion; glucose intolerance; blood biomarkers; blast overpressure
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Glucose Intolerance

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood plasma to identify blood biomarkers for blast exposure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Repetitive blast exposure has been shown to lead to more severe neurobehavioral impairments versus a single exposure. Blast-induced Traumatic Brain Injury (TBI) can lead to short- and long-term adverse outcomes Even mild brain injuries can impair neurocognitive performance, and repeated injuries can amplify negative outcomes.

Service members with repeated exposure to low-level blasts as a necessary part of their job or training display altered neural activity during a memory task that is paralleled by a reduction in accuracy on neurocognitive memory tasks. As a result, it is important to monitor service members that are exposed to multiple blast-generated mTBIs to allow the earliest identification of acute or chronic brain and body insult and provide individualized measures of time to recovery. While TBI is clinically diagnosable, the methods of diagnosis have up to now been typically expensive and immobile, and treatments and interventions sparse. The investigators will conduct a longitudinal assessment of mTBI brain biomarkers by collecting repeated measures of FDA approved mTBI brain injury biomarkers, correlated with sound and blast exposure, as well as continuous monitoring through smart watches (activity, sleep, biometrics, calorie expenditure, balance) and analyte data through analyte sensors (glucose, lactate, ketones). Study data will be organized into categories and presented to participants daily within the application and will be securely stored within the application. At the completion of the study, participants will be provided with the study data digitally within the mobile application and study data will also be provided to the credentialed unit medical provider to enable it to be ported to the participants' electronic medical record. This study will create a continuous record of blast overpressure and sound exposures and correlate those to the participants health state over the course of several 9-week courses. This will enable an assessment of individualized susceptibility to brain injury as well as providing novel data on time to recovery. The investigators hope to develop dynamic and accurate risk profiles that are individual and will lead to further understanding of how to protect participants from mTBI (mild TBI) events.

DETAILED DESCRIPTION:
Repetitive blast exposure has been shown to lead to more severe neurobehavioral impairments versus a single exposure (e.g., Gao, et al, 2017). As a result, it is important to monitor service members that are exposed to multiple blast-generated mTBIs in order to allow the earliest identification of acute or chronic brain and body insult and provide individualized measures of time to recovery. Although time to recovery and return to work decisions are critical to unit readiness, currently the prediction of outcome after mTBI is difficult, whether the outcome is measured by the time to recovery, the persistence of symptoms, or the development of a post-concussion syndrome (PCS).

Blast-induced TBI can lead to short- and long-term adverse outcomes. Many with TBI experience severe symptoms immediately following the physical trauma, with 26.1% reporting loss of consciousness and 22.4% losing memory of events before or after the injury . However, symptoms are varied (i.e. difficulty concentrating, compromised executive function, headache, confusion, amnesia, chronic pain, mental health conditions, etc.) and can present months or years after the injury, with as many as 53% of those who suffer from TBI experiencing symptoms a year or more post-injury). Long-term effects are serious and even increase the risk of chronic decline, such as dementia and Parkinson's Disease. While TBI is clinically diagnosable, the methods of diagnosis have up to now been typically expensive and immobile, and treatments and interventions sparse.

The investigators hope to learn whether daily continuous and long-term information about the physical and mental status of warfighters that is collected by wearable sensors and a mobile app can accurately monitor and predict physical and mental performance, as well as to increase warfighter self-knowledge and personal awareness on the best methods to monitor and maximize physical and mental performance. This research is being funded by the Defense Health Agency through the Congressionally Directed Medical Research Programs (CDMRP).

Participants will participate in the study for 9 weeks to 18 months during classes which they instruct. They will be asked to complete baseline surveys on the app related to demographics, personality, psychology, lifestyle, and brain function. The research mobile app is the main hub of the study and will collect data from wearable sensors (i.e. the Apple Watch) in the research study, as well as have surveys to fill out and other resources such as information on nutrition, sleep, and meditation. They may also be asked to complete daily and weekly surveys during the study. At the end of the study, they will be given additional end-of-study surveys via the mobile app, which may include surveys about experience with the wearable sensors and the mobile app, as well as other follow-up surveys.

Wearables: The Apple Watch will collect activity data including heart rate, daily steps total, estimated energy expenditure, distance moved, minutes of activity, and sleep, synched with the research mobile app and stored in a database for research analysis by the research team

Participants will be offered the continuous glucose monitor (CGM) which will collect data on glucose levels.

Blood will be drawn to test for blood biomarkers (UCH-L1 and GFAP) of blast exposure 2 times per week during most of the 9-week duration of a training class. The only exception will be during week 5 of the class, where the preponderance of blast overpressure is experienced by the cadre during breaching training. During week 5, blood will be drawn 2 times per day.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion in the study is limited to instructors of the Special Forces Advanced Reconnaissance Target Analysis and Exploitation Techniques Course (SFARTAETC) at Range 37, D Co. 2nd BN / 2nd SWTG(A) at Fort Bragg, NC.

Exclusion Criteria:

* Must be 18 yo or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Instructors of the Special Forces Advanced Reconnaissance Target Analysis and Exploitation Techniques Course (SFARTAETC) at Range 37, D Co. 2nd BN / 2nd SWTG(A) at Fort Bragg, NC.
  All participants will be employees of the Army, but they will range from Active Duty Service Members to civilian Governments employees to Contractors. All will be instructing soldiers in the SFARTAETC training course.
  All SFARTAETC instructors will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Blood Biomarkers and blast exposure | 18 months
  Determine if repeated measures of FDA approved mTBI brain injury biomarkers (for concussive injury) are correlated with sound and blast exposure. Measures of blood biomarkers, ubiquitin C-terminal hydrolase-L1 (UCH-L1) and glial fibrillary acidic protein (GFAP), will be taken to determine if they are elevated after acute or chronic blast exposure as measured with dosimeters and blast gauges.
Blood Biomarkers and neurophysiologic metrics | 18 months
  Determine if repeated measures of FDA approved mTBI brain injury biomarkers (for concussive injury) are correlated with neurophysiologic metrics. Measures of blood biomarkers, ubiquitin C-terminal hydrolase-L1 (UCH-L1) and glial fibrillary acidic protein (GFAP), will be taken to determine if they are elevated in correlation with neurophysiologic metrics such as heart rate, HRV, respiration, sleep and activity.
Blood Biomarkers and psychologic metrics | 18 months
  Determine if repeated measures of FDA approved mTBI brain injury biomarkers (for concussive injury) are correlated with psychologic metrics. Measures of blood biomarkers, ubiquitin C-terminal hydrolase-L1 (UCH-L1) and glial fibrillary acidic protein (GFAP), will be taken to determine if they are elevated in correlation with psychologic measures such as depression, PTSD, cognitive changes, and post-concussive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Ft. Bragg, Fort Bragg, North Carolina, United States